CLINICAL TRIAL: NCT05182021
Title: The Effect of Advanced Maternal Age on Pregnancy Outcomes: A Prospective Study
Brief Title: Pregnancy Outcomes on Advanced Maternal Age
Acronym: AMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MS.21.06.1542
Record Dates: First submitted 2021-10-13; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-10

CONDITIONS: Advanced Maternal Age Pregnancy
Keywords: Advanced maternal age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: The case group represented by 50 primigravida women aged 35 y or more during their pregnancy or at the time of delivery
- Control group: The control group represented by 50 primigravida women aged 20 y : 34 y during their pregnancy or at the time of delivery

SUMMARY:
A prospective observational study of pregnancy outcomes at advanced maternal age among primigravida which include maternal ,fetal, obstetric and perinatal outcomes

DETAILED DESCRIPTION:
The investigator will have 2 groups of primigravida , the first group will be presented by 50 women aged 35 y or more and the second group will be presented by 50 women aged 20 y to 34 y The first group will be also divided into 2 subgroups : group (1A ) aged 35 y to 40 y and group (1B) aged above 40 y The investigator will compare the outcomes between the two group , also comparing the outcomes between women with spontaneous pregnancy and those using ART ( Assisted Reproductive Technology ) The participants will undergo routine investigations at the first antenatal visit and a monthly ultrasound examination until delivery The participants will be screened for gestational diabetes mellitus using oral glucose tolerance test between 24 :34 weeks of pregnancy The participants will be screened for gestational hypertension after 20 weeks of pregnancy Obstetric outcomes will be recorded regarding pregnancy induced hypertension, gestational diabetes mellitus , anemia, antepartum hemorrhage, obstetric shock and intrapartum hemorrhage Maternal outcomes will be recorded regarding mode of delivery ,time of delivery ,preterm labor ,obstructed labor and prolonged labor Fetal outcomes will be recorded regarding congenital malformation ,intra uterine growth retardation ,intra uterine fetal death and still birth Perinatal outcomes will be recorded regarded birth weight ,birth asphyxia , neonatal hypoglycemia ,hyperbilirubinemia and ICU admission

ELIGIBILITY:
Inclusion Criteria:

* all primigravida women aged 20 to 34 years in control group and aged 35years or more in case group who seeking for antenatal care in mansoura university hospital and who accept study protocol

Exclusion Criteria:

* multipara
* women aged less than 20 years
* women with any medical disorder ( anti phospholipid syndrome , chronic hypertension ,Diabetes, autoimmune disease and thrombosis embolic disease )

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: The control group will be presented by 50 women aged 20-34 years during their pregnancy and the case group will be presented by 50 women aged 35 years or more during their pregnancy or at the time of delivery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the Obstetric outcomes as Gestational diabetes mellitus between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Gestational diabetes mellitus by using oral glucose tolerance test between 24 : 28 weeks of pregnancy (in mg/dl),
Comparing the Obstetric outcomes as Anemia between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Detecting Anemia by measuring hemoglobin level (in gm/dl).
Comparing the Obstetric outcomes as Oligohydramnios or polyhydramnios between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Detected by measuring (amniotic fluid index in cm) by ultrasound.
Comparing the Maternal outcomes as Preterm labor between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Preterm labor before 37 w of pregnancy calculated from last menstrual period.
Comparing the Fetal outcomes of pregnancy between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Fetal outcomes include:
  - Congenital malformation & Intra uterine fetal death (detected by anomaly scan).
Comparing the Perinatal outcomes as Birth weight between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Birth weight (in gm).
Comparing the Neonatal hypoglycemia between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Detected by measuring neonatal blood glucose level (mg/dl).
Comparing the Neonatal outcomes of pregnancy between the young and the elderly group | Between June 2021 to June 2022 and may be extended if needed
  Include:
  * APGAR score system.
  * Neonatal intensive care unit admission

SECONDARY OUTCOMES:
Comparing the Obstetric outcomes as Gestational diabetes mellitus between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Gestational diabetes mellitus by using oral glucose tolerance test between 24 : 28 weeks of pregnancy (in mg/dl),
Comparing the Obstetric outcomes as Anemia between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Detected by measuring hemoglobin level (in gm/dl).
Comparing the Obstetric outcomes as Oligohydramnios or polyhydramnios between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Oligohydramnios or polyhydramnios by measuring (amniotic fluid index in cm) by ultrasound.
Comparing the Maternal outcomes of pregnancy between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Preterm labor before 37 w of pregnancy calculated from last menstrual period.
Comparing the Fetal outcomes of pregnancy between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Congenital malformation & Intra uterine fetal death (detected by anomaly scan).
Comparing the Perinatal outcomes as Birth weight between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Birth weight (in gm).
Comparing the Neonatal hypoglycemia of pregnancy between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Neonatal hypoglycemia by measure neonatal blood glucose level (mg/dl).
Comparing the Neonatal outcomes of pregnancy between women with spontaneous pregnancy and those using Assisted Reproductive Technique | Between June 2021 to June 2022 and may be extended if needed
  Include:
  * APGAR score system.
  * Neonatal intensive care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Rana magdy ibrahim El gharbawy, Principal Investigator — Obstetric and Gynecology department at mansoura university hospital
Locations (1):
- Mansoura university hospital, Al Mansurah, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT05182021/Prot_SAP_000.pdf